CLINICAL TRIAL: NCT06821204
Title: Detection of Pathogenic Bacteria in Make-up Tools and Evaluation of Hygiene Education Effectiveness
Brief Title: Detection of Pathogenic Bacteria in Make-up Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Duygu Akçay, Assistant Professor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UFUKU-HSH-DA-01
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Health Education
Keywords: Makeup Tools; Pathogenic Bacteria; Hygiene Education
MeSH Terms: conditions — Health Education | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two groups with a control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will not be informed about group assignments and will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healt Education Group (Active Comparator): Participants will be given one session (40 minutes) of training on the definition and importance of hygiene, the rules and importance of hand washing, the importance of cleaning make-up materials, which method, material and how often they should be cleaned, and the health risks that may occur if they are not cleaned.
  Interventions: Other: Health education group
- Control group (Sham Comparator): No intervention will be applied to participants in this group.
  Interventions: Other: control group

INTERVENTIONS:
Other: Health education group — Participants will be given one session (40 minutes) of training on the definition and importance of hygiene, the rules and importance of hand washing, the importance of cleaning make-up materials, which method, material and how often they should be cleaned, and the health risks that may occur if they are not cleaned.
  Arms: Healt Education Group
Other: control group — No intervention will be applied to participants in this group.
  Arms: Control group

SUMMARY:
In addition to collecting product residues, dirt and oil, makeup products can damage the skin and cause infection as they are a breeding ground for bacteria. Studies investigating the microbiological contamination of makeup applicators have shown that makeup sponges and brushes are a means of transmitting pathogens. Other studies have determined that positive isolates are detected in almost every device taken from makeup tools. In order to draw attention to the source of infection that is not widely known by the public and to instill correct hygiene habits, this study aims to detect pathogenic bacteria in makeup tools used by university students and to evaluate the effectiveness of the hygiene training provided.

DETAILED DESCRIPTION:
Makeup does a good job of improving the appearance of women. However, many women do not know that makeup can be a health hazard because it contains bacteria and can spread infection. In addition to collecting product residue, dirt, and oil, makeup products can damage the skin and cause infection because they are a breeding ground for bacteria. Cosmetic contamination leads to various types of infections, ranging from mild to serious.

Studies investigating the microbiological contamination of used makeup applicators have shown that makeup sponges and brushes are a vehicle for pathogen transmission. Other studies have determined that Staphylococcus aureus grows as the dominant bacteria in makeup tools and that positive isolates are detected in almost every device taken. The American Academy of Dermatology recommends washing your makeup brushes every 7 to 10 days to protect your skin and kill any harmful bacteria left on your makeup brushes.

Infectious diseases are still a major public health problem, especially in developing countries. Therefore, it is important for people to adopt proper hygiene habits, especially hand washing, to prevent infection. In order to draw attention to a source of infection that is not widely known by the public and to instill correct hygiene habits, this study aims to detect pathogenic bacteria in make-up tools used by university students and to evaluate the effectiveness of the hygiene education provided.

ELIGIBILITY:
Inclusion Criteria:

* Being registered at Ufuk University School of Nursing,
* Being over 18 and under 30
* Being female,
* Having make-up tools,
* Being volunteer to participate in the research.

Exclusion Criteria:

* Being male,
* Not having make-up tools,
* Giving up participating in the research,
* Under 18 years old, over 30 years old

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Hygiene Control Kit | two weeks
  A kit designed to perform microbiological analysis in a practical way will be used to reveal the microorganism density and pathogenic microorganism presence in the make-up tools swab sample. The Hygiene Control Kit (Hytech Slide product) is in compliance with the ISO 18593:2004 Standard.
  The kit is a product that can perform analysis with medium contact from all surfaces for microbiological analysis. It is possible to take samples from all surfaces, personnel, equipment, solid and liquid. Thanks to its 90-degree bendable structure, the medium comes into contact with the surface even on difficult, inclined and narrow surfaces. E.coli and S.Aureus colonies will be counted after incubation.

SECONDARY OUTCOMES:
Individual information form | two weeks
  The individual information form was developed based on relevant literature. The form includes 22 questions to determine the frequency and method of infection, hand washing, makeup use and cleaning of makeup tools, frequency of changing, and sharing with someone else.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akçay, Asst. Prof., Principal Investigator — Ufuk University; Aslı Genç, Asst. Prof., Principal Investigator — Ufuk University; Nedim Sultan, Prof.Dr., Principal Investigator — Ufuk University
Locations (1):
- Ufuk University, Balgat, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No